CLINICAL TRIAL: NCT03076970
Title: A Randomized, Double-Blind, Three Period, Cross-Over Study to Evaluate the Effect of Single Oral Doses of Lasmiditan When Coadministered With Single Oral Doses of Sumatriptan (Imitrex) in Healthy Male and Female Subjects
Brief Title: Effect of Single Oral Doses of Lasmiditan When Coadministered With Single Oral Doses of Sumatriptan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: SNBL Clinical Pharmacology Center, Inc. (Industry); CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16885; COL MIG-118 (Other: CoLucid Pharmaceuticals); H8H-CD-LAHI (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lasmiditan 200 mg (Experimental): single oral tablet
  Interventions: Drug: lasmiditan 200 mg; Drug: matching placebo
- Sumatriptan 100 mg (Active Comparator): single oral tablet
  Interventions: Drug: Sumatriptan; Drug: matching placebo
- Combination of lasmiditan and sumatriptan (Experimental): single oral tablet of each
  Interventions: Drug: lasmiditan 200 mg; Drug: Sumatriptan

INTERVENTIONS:
Drug: lasmiditan 200 mg — drug including single placebo tablet
  Other Names: LY573144
  Arms: Combination of lasmiditan and sumatriptan; Lasmiditan 200 mg
Drug: Sumatriptan — drug including single placebo tablet
  Arms: Combination of lasmiditan and sumatriptan; Sumatriptan 100 mg
Drug: matching placebo — single oral tablet -given with single lasmiditan tablet and with single sumatriptan tablet.
  Arms: Lasmiditan 200 mg; Sumatriptan 100 mg

SUMMARY:
This is a randomized, double-blind, three-period, cross-over study to investigate the effect of sumatriptan (Imitrex) 100 mg on the pharmacodynamics and pharmacokinetics of lasmiditan 200 mg.

DETAILED DESCRIPTION:
This is a randomized, double-blind, three-period, cross-over study to investigate the effect of single doses of sumatriptan (Imitrex) 100 mg on the pharmacodynamics of single doses of lasmiditan 200 mg. The study will last approximately 6 weeks including up to 3 weeks for screening and 22 days on study. Screening will be conducted within approximately 21 days of the first dose of study medication. Each dosing period will last 3 days (Day 1, Day 1, and Day 2). A wash-out period of 6 days will take place between each dose. The End of Study Visit (EoS) will take place 5 (+/- 2) days after the third dosing period is completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60 years, inclusive.
* Able and willing to give written informed consent.
* Body mass index (BMI) between 18 and 32 kilograms per square meter (kg/m²), inclusive.
* Participants must be able to refrain from consuming xanthine, quinine and caffeine containing beverages, and must refrain from prolonged intensive physical exercise during the study (from 72 hours prior to dosing until the end of study).
* Women must be:

  * not pregnant
  * not breast-feeding
  * not planning to become pregnant during the study
* All females must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in on Day -1 of each period. All women must agree to use an adequate method of contraception during the study and for 30 days following the end-of-study.
* Male participants must agree to utilize a highly effective method of contraception (condom plus spermicide) during heterosexual intercourse from clinic admission until 30 days following the end of study.
* Male participants must agree to refrain from sperm donation from clinic admission until at least 30 days following the end of study.
* Participants must be able to swallow multiple pills simultaneously.
* Participants must be able to understand the requirements of the study and must be willing to comply with the requirements of the study.

Exclusion Criteria:

* Any medical condition, clinical laboratory test or other reason which in the judgment of the Investigator or designee makes the participant unsuitable for the study.
* Any clinically significant abnormalities (as determined by the Principal Investigator or designee) in hematology, blood chemistry and/or urinalysis lab tests at screening or at Period 1 D-1.
* Known hypersensitivity to lasmiditan, sumatriptan (Imitrex), or to any excipient of lasmiditan or sumatriptan (Imitrex) oral tablets.
* Use of any prescription medication, including monoamine oxidase A (MAO-A) inhibitors and other drugs associated with serotonin syndrome, within 14 days prior to dosing (except hormonal contraceptives) except for 5-HT1 (serotonin) agonists and selective serotonin reuptake inhibitors.
* History, symptoms, or signs of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes including but not limited to angina pectoris, myocardial infarction, silent myocardial ischemia (Ischemic cardiac syndromes), stroke, transient ischemic attacks (cerebrovascular syndromes), and ischemic bowel disease (peripheral vascular disease).
* History, symptoms, or signs of vasospastic coronary artery disease.
* History, symptoms, or signs of arrhythmia or Wolff Parkinson White (WPW) syndrome that could affect the participant's safety in the opinion of the Investigator or designee.
* History, symptoms, or signs of severe hepatic impairment.
* History, symptoms, or signs of diabetes.
* History within the previous 3 years or current evidence of abuse (according to Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition [DSM-IV] criteria) of any drug, prescription or illicit, or alcohol; a positive urine screen for drugs of abuse or breathalyzer alcohol test.
* Positive urinary test for drugs of abuse and/or alcohol breath test at Screening and/or at check-in on Day -1 of each Period. Cotinine will be included at screening only.
* History of orthostatic hypotension with or without syncope.
* Supine systolic blood pressure (BP) > 135 millimeters of mercury (mmHg), diastolic BP > 85 mm Hg, respiratory rate >20 breaths per minute, pulse >90 beats per minute, or temperature >37.5º at Screening. Low values on any vital sign measurement will be assessed at the discretion of the Investigator or designee. For orthostatic vital signs, any decrease in systolic and/or diastolic blood pressure great than 20 mmHg. Any other changes will be assessed at the discretion of the Investigator or designee.
* Electrocardiogram (ECG) changes including QT interval prolongation and congenital long QT syndrome.
* Electrolyte abnormalities (e.g., hypokalemia or hypomagnesemia), congestive heart failure, or other medicinal products that lead to QT prolongation.
* Any clinically significant alanine aminotransferase (ALT), alkaline phosphatase (AP), aspartate aminotransferase (AST), or bilirubin abnormalities judged by the Investigator or designee at Screening.
* Treatment with centrally active drugs or those affecting peripheral cholinergic transmission within 3 months of study entry.
* Consumption of grapefruit, grapefruit juice, Seville oranges, Seville orange juice, or beverages containing any of these juices or consumption of members of the mustard green family (including kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard (i.e. seeds, greens, spice or the condiment)) within 72 hours of dosing.
* Tobacco or nicotine users except participants who stopped using tobacco or nicotine 1 year or more before signing the informed consent.
* Participant is at imminent risk of suicide or had a suicide attempt within 6 months prior to screening .
* Participation in any clinical trial of an experimental drug or device in the previous 30 days.
* Positive Hepatitis C antibody, Hepatitis B surface antigen, or positive human immunodeficiency virus (HIV) antibody.
* Participants who donated plasma in the 7 days or blood in the 3 months - Participants with an inability to communicate well with the Investigator or designee and study staff (i.e., language problem, poor mental development or impaired cerebral function).
* Inability to fast or consume the food provided in the study.
* Relatives of or staff directly reporting to the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- SNBL Clinical Pharmacology Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with three study periods, participants were randomly allocated to one of six treatment sequences: ABC, ACB, BAC, BCA, CAB or CBA as per the dosing sequence in each period with 6 days washout period.
Groups:
- Sequence ABC: Single oral doses of lasmiditan co-administered with single oral doses of sumatriptan (Imitrex) in the following sequence:
  Period 1 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo. Period 2 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo. Period 3 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
- Sequence ACB: Single oral doses of lasmiditan co-administered with single oral doses of Sumatriptan (Imitrex) in the following sequence:
  Period 1 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo. Period 2 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
  Period 3 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo.
- Sequence BCA: Single oral doses of lasmiditan co-administered with single oral doses of sumatriptan (Imitrex) in the following sequence:
  Period 1 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo. Period 2 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
  Period 3 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo.
- Sequence BAC: Single oral doses of lasmiditan co-administered with single oral doses of sumatriptan (Imitrex) in the following sequence:
  Period 1 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo. Period 2 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo. Period 3 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
- Sequence CAB: Single oral doses of lasmiditan co-administered with single oral doses of sumatriptan (Imitrex) in the following sequence:
  Period 1 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
  Period 2 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo. Period 3 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo.
- Sequence CBA: Single oral doses of lasmiditan co-administered with single oral doses of Sumatriptan (Imitrex) in the following sequence:
  Period 1 (C): lasmiditan 200 mg co-administered with sumatriptan (Imitrex) 100 mg.
  Period 2 (B): sumatriptan (Imitrex) 100 mg + lasmiditan 200 mg placebo. Period 3 (A): lasmiditan 200 mg + lasmiditan 200 mg placebo.
Period: Period 1
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 7 | 7
Received at Least 1 Dose of Study Drug | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 7 | 7 | 7 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Failure to meet I/E criteria | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period 3
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 7 | 7 | 7 | 7 | 5 | 6
Completed | 7 | 7 | 7 | 7 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug (lasmiditan or sumatriptan).
Groups:
- Overall: Single oral doses of Lasmiditan 200 mg, lasmiditan 200 mg placebo and sumatriptan (Imitrex) 200 mg administered as per the dosing sequence in each period.
Arm/Group | Overall
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 11
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in Vital Signs: Systolic Blood Pressure
Description: Vital signs were measured in semi-supine position after 5 minutes rest. Serial vital signs assessed when lasmiditan is administered alone and when sumatriptan is administered alone compared to when lasmiditan and sumatriptan are administered together.
Time Frame: Pre-dose, 24 hours post-dose
Population: All participants who received at least one dose of study drug (lasmiditan or sumatriptan) and have completed at least one treatment period.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Lasmiditan 200 mg: Participants received single oral tablet of lasmiditan 200 mg with lasmiditan 200 mg placebo.
- Sumatriptan 100 mg: Participants received single oral tablet of sumatriptan 100 mg with lasmiditan 200 mg placebo.
- Combination of Lasmiditan and Sumatriptan: Participants received single oral tablet of lasmiditan 200 mg with sumatriptan 100 mg.
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
millimeters of mercury (mmHg) | 0.6 (7.03) | -2.3 (12.88) | -0.1 (8.22)

2. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in Vital Signs: Diastolic Blood Pressure
Description: as for outcome 1
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
mmHg | -1.3 (6.33) | -1.1 (7.53) | 0.6 (6.14)

3. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in Vital Signs: Pulse Rate
Description: as for outcome 1
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
beats/min | -2.5 (9.75) | -1.0 (9.51) | 1.8 (7.46)

4. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in Vital Signs: Temperature
Description: as for outcome 1
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
Celsius (C) | 0.0 (0.51) | -0.0 (0.41) | -0.1 (0.54)

5. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in Vital Signs: Respiratory Rate
Description: as for outcome 1
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
breaths/min | 0.2 (2.35) | 0.2 (1.95) | 0.7 (1.69)

6. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: Heart Rate
Description: A standard, digital 12-lead ECG with a 10-second rhythm strip was used to assess cardiac function after participants have been at least 5 minutes supine. Serial ECGs collected when lasmiditan administered alone and when sumatriptan is administered alone compared to when lasmiditan and sumatriptan are administered together.
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
beats/min | -0.8 (6.49) | -1.3 (4.99) | 0.4 (5.75)

7. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: Summary (Mean) PR Duration
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
milliseconds (msec) | -4.5 (10.79) | -2.5 (10.85) | -1.6 (11.22)

8. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: Summary (Mean) QRS Duration
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
msec | -0.5 (4.67) | -1.7 (4.44) | -0.6 (4.83)

9. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: QTcB - Bazett's Correction Formula
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
msec | -2.7 (14.07) | -3.3 (11.27) | 1.6 (11.64)

10. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: QTcF - Fridericia's Correction Formula
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
msec | -1.8 (9.48) | -2.0 (8.91) | 1.3 (8.54)

11. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: Summary (Mean) QT Duration
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
msec | 0.1 (12.19) | 1.0 (11.84) | 0.6 (12.44)

12. Primary Outcome: Pharmacodynamics- Change From Pre-dose to 24 Hours in ECGs: Summary (Mean) RR Duration
Description: as for outcome 6
Time Frame: Pre-dose, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
msec | 14.1 (91.17) | 24.2 (77.23) | -4.1 (84.28)

13. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety assessed from time of consent through end of study. A summary of all reported serious adverse events (SAE) and other adverse events regardless of causality are provided in the adverse events module of this record.
Time Frame: Up to 6 weeks
Population: All participants who received at least one dose of study drug (lasmiditan or sumatriptan).
Measure: Count of Participants; unit: Participants
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 40 | 42
Participants
  Adverse Events (AEs) | 24 | 16 | 28
  Serious Adverse Events (SAEs) | 0 | 0 | 0

14. Secondary Outcome: Pharmacokinetics - Cmax
Description: Maximum plasma concentration of lasmiditan alone compared to lasmiditan in combination with sumatriptan.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 30 hours following the dose at time 0 in each dosing period
Population: All participants who completed at least one treatment period without any protocol violations, who have evaluable plasma concentration data for lasmiditan and/or sumatriptan (Imitrex), and for whom at least a subset of the designated PK parameters can be determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lasmiditan Alone: Participants received single oral tablet of lasmiditan 200 mg.
Arm/Group | Lasmiditan Alone | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 42
nanogram per milliliter (ng/mL) | 268 (40) | 238 (37)

15. Secondary Outcome: Pharmacokinetics - AUC0-t
Description: Area under the plasma concentration versus time curve from time 0 to the time t of the last quantifiable concentration, calculated by means of the mixed log-linear trapezoidal rule of lasmiditan alone compare to lasmiditan in combination with sumatriptan.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Lasmiditan Alone | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 42
nanogram*hour per milliliter (ng*h/mL) | 1730 (35) | 1650 (35)

16. Secondary Outcome: Pharmacokinetics - Tmax
Description: Time to maximum plasma concentration of lasmiditan alone compared to lasmiditan in combination with sumatriptan.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Full Range); unit: hour
Arm/Group | Lasmiditan Alone | Combination of Lasmiditan and Sumatriptan
Number analyzed (Participants) | 41 | 42
hour | 2.00 [1 to 4] | 3.00 [1 to 6]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: All participants who received at least one dose of study drug (lasmiditan or sumatriptan).
Arm/Group | Lasmiditan 200 mg | Sumatriptan 100 mg | Combination of Lasmiditan and Sumatriptan
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 24/41 | 16/40 | 28/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lasmiditan 200 mg (N=41) | Sumatriptan 100 mg (N=40) | Combination of Lasmiditan and Sumatriptan (N=42)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (4)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 14 (14) | 3 (3) | 12 (12)
Headache (Nervous system disorders) | 2 (3) | 7 (7) | 8 (8)
Hypersomnia (Nervous system disorders) | 9 (9) | 4 (4) | 16 (16)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
Euphoric mood (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03076970/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03076970/SAP_001.pdf